CLINICAL TRIAL: NCT07282106
Title: Effect of Transcutaneous Auricular Stimulation of the Vagus Nerve on Functional Connectivity in the Brain at Rest: fNIRS Study in Chronic Post-stroke Subjects and Healthy Subjects
Brief Title: Effect of Transcutaneous Auricular Stimulation of the Vagus Nerve on Functional Connectivity in the Brain at Rest
Acronym: COVAGNIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Les Trois Soleils (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-A01694-45; 25.03521.000408 (Registry Identifier: SI RIPH 2G)
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Stroke Patients
Keywords: fNIRS; taVNS; stroke; functional brain connectivity; resting state; healthy people
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active taVNS arm (Experimental): Transcutaneous Auricular Vagus Nerve Stimulation (taVNS): Delivery of low-intensity electrical impulses to the outer ear (concha and tragus) to stimulate the auricular branch of the vagus nerve.
  Interventions: Device: Active taVNS arm
- Sham Control arm (Sham Comparator): Simulated/Placebo Stimulation (Sham): Application of the device without delivering an active electrical current, serving as the necessary control condition.
  Interventions: Device: Sham Control arm

INTERVENTIONS:
Device: Active taVNS arm — Transcutaneous Auricular Vagus Nerve Stimulation (taVNS): Delivery of low-intensity electrical impulses to the outer ear (concha and tragus) to stimulate the auricular branch of the vagus nerve.
  Arms: Active taVNS arm
Device: Sham Control arm — Simulated/Placebo Stimulation (Sham): Application of the device without delivering an active electrical current, serving as the necessary control condition.
  Arms: Sham Control arm

SUMMARY:
The goal of this clinical trial is to study the effect of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on resting-state brain functional connectivity. The study will assess this effect using functional Near-Infrared Spectroscopy (fNIRS) in both chronic post-stroke patients and healthy subjects.

The main questions it aims to answer are:

Does taVNS affect resting-state functional connectivity (measured by fNIRS) in chronic post-stroke patients?

Does taVNS affect resting-state functional connectivity (measured by fNIRS) in healthy subjects?

Are there differences in the effect of taVNS on functional connectivity between the post-stroke group and the healthy group?

Researchers will compare the effect of active taVNS (real stimulation) to a sham stimulation (control) to evaluate its specific impact on the brain's functional networks.

ELIGIBILITY:
Inclusion Criteria for post-stroke participant:

* age 18 or older
* Right-handed participant;
* Hemiparesis in the chronic phase (>6 months post-stroke)
* Participant who has agreed to sign an informed consent form;
* Participant who is affiliated with social security.

Inclusion Criteria for healthy participant:

* age 18 or older
* Right-handed participant;
* Participant who has agreed to sign an informed consent form;
* Participant who is affiliated with social security.

Exclusion Criteria for post-stroke participant:

* Allergy to neoprene (the material used to make the fNIRS cap);
* Hair volume preventing the cap from being put on and/or access to the scalp;
* Cognitive impairment making it impossible to participate in the study;
* Phasic disorders preventing understanding of instructions and effective communication;
* Pregnant or breastfeeding women;
* Persons under legal protection

Exclusion Criteria for post-stroke participant:

* Allergy to neoprene (the material used to make the fNIRS cap);
* Hair volume preventing the cap from being put on and/or access to the scalp;
* Pregnant or breastfeeding women;
* Persons under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Resting-State Functional Connectivity | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Les Trois Soleils, Boissise-le-Roi, France

IPD SHARING:
Plan to Share IPD: No